CLINICAL TRIAL: NCT02551809
Title: A Randomized, Double-blind, Placebo-controlled, 3-arm Parallel-group, Multicenter, Phase IIa Study to Evaluate the Safety, Tolerability, Immunogenicity, and Efficacy of UBITh® AD Immunotherapeutic Vaccine (UB-311) in Patients With Mild Alzheimer's Disease
Brief Title: Evaluate the Safety, Tolerability, Immunogenicity and Efficacy of UB-311 in Mild Alzheimer's Disease (AD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Neuroscience Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V203-AD
Record Dates: First submitted 2015-09-10; First posted 2015-09-16 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 3 priming doses followed by 4 boosters (Experimental): Subjects will receive 7 doses of UB-311.
  Interventions: Biological: UB-311
- 3 priming doses followed by 2 boosters (Experimental): Subjects will receive 5 doses of UB-311 and 2 doses of placebo.
  Interventions: Biological: UB-311; Drug: Placebo
- Placebo (Placebo Comparator): Subjects will receive 7 doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: UB-311 — Intramuscular injection
  Arms: 3 priming doses followed by 2 boosters; 3 priming doses followed by 4 boosters
Drug: Placebo — Intramuscular injection
  Arms: 3 priming doses followed by 2 boosters; Placebo

SUMMARY:
The purpose of this Phase IIa study is to determine whether the AD Immunotherapeutic Vaccine (UB-311), targeting the amyloid beta peptide (N-terminal amino acids, 1-14), is safe and immunogenic in mild AD patients. In addition, the efficacy profiles will be evaluated as the secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild Alzheimer's Disease
* Mini-Mental State Examination (MMSE) scores between 20 and 26 (inclusive)
* Clinical dementia rating (CDR) scores of 0.5 or 1
* Other inclusion criteria apply

Exclusion Criteria:

* Clinically significant neurological disease other than Alzheimer's disease
* Major psychiatric disorder
* Severe systemic disease
* Serious adverse reactions to any vaccine
* Other exclusion criteria apply

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital (KS-CGMH), Kaohsiung City
  - National Taiwan University Hospital (NTUH), Taipei
  - Taipei Veterans General Hospital (TVGH), Taipei
  - Linkou Chang Gung Memorial Hospital (LK-CGMH), Taoyuan District

REFERENCES:
- [Derived] Yu HJ, Dickson SP, Wang PN, Chiu MJ, Huang CC, Chang CC, Liu H, Hendrix SB, Dodart JC, Verma A, Wang CY, Cummings J. Safety, tolerability, immunogenicity, and efficacy of UB-311 in participants with mild Alzheimer's disease: a randomised, double-blind, placebo-controlled, phase 2a study. EBioMedicine. 2023 Aug;94:104665. doi: 10.1016/j.ebiom.2023.104665. Epub 2023 Jun 29. PMID 37392597
- [Derived] Wang CY, Wang PN, Chiu MJ, Finstad CL, Lin F, Lynn S, Tai YH, De Fang X, Zhao K, Hung CH, Tseng Y, Peng WJ, Wang J, Yu CC, Kuo BS, Frohna PA. UB-311, a novel UBITh(R) amyloid beta peptide vaccine for mild Alzheimer's disease. Alzheimers Dement (N Y). 2017 Apr 14;3(2):262-272. doi: 10.1016/j.trci.2017.03.005. eCollection 2017 Jun. PMID 29067332
- See also: Site-specific UBITh amyloid-beta vaccine for immunotherapy of Alzheimer's disease. — http://www.ncbi.nlm.nih.gov/pubmed/17287052?dopt=Abstract

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3 Priming Doses Followed by 4 Boosters | 3 Priming Doses Followed by 2 Boosters | Placebo
Started | 14 | 15 | 14
Completed | 14 | 14 | 13
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Priming Doses Followed by 4 Boosters | 3 Priming Doses Followed by 2 Boosters | Placebo | Total
Number analyzed (Participants) | 14 | 15 | 14 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (6.81) | 72.5 (6.79) | 72.0 (7.62) | 72.6 (6.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 11 | 32
  Male | 3 | 5 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 14 | 15 | 14 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
APOE4 carrier [Count of Participants; unit: Participants] | 10 | 12 | 13 | 35

OUTCOME MEASURES:

1. Primary Outcome: Tolerability and Safety Profile of UB-311 Assessed Via Recording of Number of Participants With Adverse Events
Description: Safety endpoints include local tolerability at the injection site, amyloid-related imaging abnormalities, vital signs, physical examination, 12-lead ECG, laboratory tests and other AEs and SAEs.
Time Frame: 78 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Priming Doses Followed by 4 Boosters | 3 Priming Doses Followed by 2 Boosters | Placebo
Number analyzed (Participants) | 14 | 15 | 14
Participants | 10 | 13 | 13

ADVERSE EVENTS:
Time Frame: 78 weeks
Arm/Group | 3 Priming Doses Followed by 4 Boosters | 3 Priming Doses Followed by 2 Boosters | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14 | 3/15 | 2/14
Other Adverse Events (participants affected / at risk) | 4/14 | 6/15 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 Priming Doses Followed by 4 Boosters (N=14) | 3 Priming Doses Followed by 2 Boosters (N=15) | Placebo (N=14)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 Priming Doses Followed by 4 Boosters (N=14) | 3 Priming Doses Followed by 2 Boosters (N=15) | Placebo (N=14)
Injection site pain (General disorders) | 0 (0) | 4 (4) | 3 (10)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 2 (3)
Weight decreased (Investigations) | 2 (2) | 1 (2) | 1 (1)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 2 (5) | 2 (3) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site PIs must jointly publish results, unless permission is granted by Sponsor. If a joint publication is not done within 12 months after trial completion and database lock, then the site may publish its own results; provided that, a) Sponsor has 45 business days to review the proposed publication; b) the PI must delete any confidential information identified by Sponsor; and c) the PI must delay disclosure for 1 year if a patent application is filed by Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT02551809/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT02551809/SAP_002.pdf